CLINICAL TRIAL: NCT03746574
Title: Achieving the Quadruple Aim by Reducing Burnout: A Randomized Trial of a Compassion Based Curriculum for Outpatient Teams
Brief Title: Achieving the Quadruple Aim by Reducing Burnout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Providence Health & Services (Other)
Responsible Party: Principal Investigator, Mark Rosenberg, MD, Director, Compassionate Care, Providence Health & Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-132
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Intervention Model Description: Randomization to intervention or control occuring at the level of clinic. All participants within a clinic are assigned to same group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Clinics (Experimental): Participants in the intervention clinics experienced a 12 session compassion curriculum intevention offered every other week for six months. Each session lasted 80 minutes and all staff at the intervention clinics were expected to participate. A total of 16 hours of experiences were provided.
  Interventions: Behavioral: Compassion Curriculum
- Control Clinics (No Intervention): Completed baseline, end of curriculum, and 6 month follow up survey. Otherwise no intervention

INTERVENTIONS:
Behavioral: Compassion Curriculum — 12 session curriculum offered every other week for six months. Each session lasted 80 minutes and all staff at the intervention clinics were expected to participate. A total of 16 hours of experiences were provided.
  Arms: Intervention Clinics

SUMMARY:
To demonstrate that a multimodal intervention can reduce burnout in a multidisciplinary primary care practice while improving other components of the Quadruple Aim including staff engagement, patient experience, productivity and quality.

DETAILED DESCRIPTION:
Recruitment

This was a randomized trial of eleven internal medicine and family medicine clinics of Providence Medical Group (PMG) in Portland Oregon. All of the clinics were non-residency clinics. The study was conducted between January 2015 and January 2016. Introductory meetings were held with leadership dyads (medical director and manager) of all 23 clinics in the Portland area to overview the curriculum and outline conditions of study participation. Expectations included: holding the curriculum sessions during usual work hours, endorsement of participation by clinic staff, and that specific individuals would be identified to facilitate sessions for the clinic. Leadership of each clinic, subsequently, discussed the curriculum with the staffs of the clinics and eleven committed to participate and were then randomized. The staffs of the intervention clinics then received the twelve session Strengthening Compassion curriculum. Four of the intervention clinics held the sessions at the beginning of the day and opened clinic 80 minutes late. One clinic held the sessions during an extended lunch hour.

Randomization and Follow-up

Eleven clinics volunteered to participate. (47.8% of eligible clinics) Five clinics were randomly selected to participate in the Strengthening Compassion curriculum and six were selected as controls.

341 individuals participated in the study, including providers, clinical, and administrative staff. The baseline survey was completed by 153 participants in the intervention clinics and 188 participants in the control clinics. 244 of the initial participants completed a survey at the end of the intervention period and 191 at 6 month follow up Participants in the intervention clinics engaged in a 12 session curriculum offered every other week for six months. Each session lasted 80 minutes and all staff at the intervention clinics were expected to participate. A total of 16 hours of experiences were provided.

Each session was facilitated by internal non-physician staff (e.g. social workers, medical assistants, nurses) recruited by clinic leadership. The facilitators received two hours of on-line training in group facilitation, mindfulness meditation, content/exercises for each session, and were provided with a detailed facilitators guide. The facilitators also received one half hour of additional training before each session via networked phone calls and were supported by on-line materials.

Study Outcomes

Outcomes were measured utilizing a fifty one question survey administered at baseline, at the end of the 6-month curriculum and at 6 months follow-up. This survey was a composite of validated surveys that measure compassion, mindfulness, burnout, clinic relations, job satisfaction, and clinical satisfaction. The Compassion component of the survey used the Santa Clara Brief Compassion Scale (SCBCS). Mindfulness was measured with the Mindful Attention Awareness Scale (MAAS). Burnout was measured with the Maslach Burnout Inventory-Human Services Survey for Medical Personnel (MBI-HSS (MP)) comprised of three sub-scales that measure emotional exhaustion, depersonalization, and personal accomplishment. Questions about caregiver roles in the clinic, clinic relations, job satisfaction, clinical satisfaction, time working in the clinic, and time working in healthcare, were derived from a previously utilized survey provided by the Center for Outcomes Research and Education of the Providence Health and Services. Data on caregiver engagement was collected in October 2015 and October 2016 via organization wide survey through Willis-Tower-Watson. Engagement and disengagement are pre-defined categories on the Willis-Tower Watson survey. Patient experience data was collected by Press Ganey as part of their standard survey process. Impact on productivity and quality were assessed from data, routinely collected, in the Providence St. Joseph Health administrative data base.

ELIGIBILITY:
Inclusion Criteria:

* All employees working in selected clinics

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Burnout Score on Maslach Burnout Inventory | Baseline, 6 Months and 12 Months
  Score on Maslach Burnout Inventory: Maslach Burnout Inventory - Human Services Survey (MBI-HSS) is a 22-item survey that covers 3 areas: Emotional exhaustion (EE), Depersonalization (DP), and Low sense of personal accomplishment (PA). There are multiple questions for each of these subscales and responses are in the form of a frequency rating scale (never, a few times a year or less, once a month or less, a few times a month, once a week, a few times a week, every day).
Change in Compassion: Score on Santa Clara Brief Compassion Scale | Baseline, 6 Months and 12 Months
  Score on Santa Clara Brief Compassion Scale: The Santa Clare Brief Compassion Scale is a brief index that assesses compassion and its link to prosocial behaviors. An example from a 'compassion for humanity' item include ""When I hear about someone (a stranger) going through a difficult time, I feel a great deal of compassion for him or her." Responses are given on a 7-point scale from "Not at all true for me" to "Very true for me."
Change in Mindfulness: Mindful Attention Awareness Score | Baseline, 6 Months and 12 Months
  Mindful Attention Awareness Score: The trait MAAS is a 15-item scale designed to assess a core characteristic of mindfulness, namely, a receptive state of mind in which attention, informed by a sensitive awareness of what is occurring in the present, simply observes what is taking place. Scored on a scale 1=almost never--> 6=almost always
Change in Intent to stay on Caregiver survey | Baseline and 12 months
  Intent to stay on Caregiver survey

SECONDARY OUTCOMES:
Change inCaregiver Engagement measured on annual Willis Tower Watson Survey | Baseline and 12 months
  Caregiver Engagement measured on annual Willis Tower Watson Survey
Change in Patient Experience on routine Press Ganey Survey | Baseline, 6 Months and 12 Months
  Patient Experience on routine Press Ganey Survey
Change in Visit per month | Baseline, 6 Months and 12 Months
  Average number of visits
Change in Panel Size | Baseline, 6 Months and 12 Months
  Panel Size per FTE
Change in Diabetes Control | Baseline, 6 Months and 12 Months
  HbA1c
Change in BP control | Baseline, 6 Months and 12 Months
  % people with blood pressure <140/80
Change in Cancer Screening Rate | Baseline, 6 Months and 12 Months
  Average of rates of screening for breast, colon, and cervical cancer

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rosenberg, MD, Principal Investigator — Providence St. Joseph

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bodenheimer T, Sinsky C. From triple to quadruple aim: care of the patient requires care of the provider. Ann Fam Med. 2014 Nov-Dec;12(6):573-6. doi: 10.1370/afm.1713. PMID 25384822
- [Background] Hall LH, Johnson J, Watt I, Tsipa A, O'Connor DB. Healthcare Staff Wellbeing, Burnout, and Patient Safety: A Systematic Review. PLoS One. 2016 Jul 8;11(7):e0159015. doi: 10.1371/journal.pone.0159015. eCollection 2016. PMID 27391946
- [Background] Salyers MP, Bonfils KA, Luther L, Firmin RL, White DA, Adams EL, Rollins AL. The Relationship Between Professional Burnout and Quality and Safety in Healthcare: A Meta-Analysis. J Gen Intern Med. 2017 Apr;32(4):475-482. doi: 10.1007/s11606-016-3886-9. Epub 2016 Oct 26. PMID 27785668
- [Background] Panagioti M, Geraghty K, Johnson J, Zhou A, Panagopoulou E, Chew-Graham C, Peters D, Hodkinson A, Riley R, Esmail A. Association Between Physician Burnout and Patient Safety, Professionalism, and Patient Satisfaction: A Systematic Review and Meta-analysis. JAMA Intern Med. 2018 Oct 1;178(10):1317-1331. doi: 10.1001/jamainternmed.2018.3713. PMID 30193239 (Retraction: PMID 32421149 JAMA Intern Med. 2020 Jul 1;180(7):931)
- [Background] West CP, Dyrbye LN, Rabatin JT, Call TG, Davidson JH, Multari A, Romanski SA, Hellyer JM, Sloan JA, Shanafelt TD. Intervention to promote physician well-being, job satisfaction, and professionalism: a randomized clinical trial. JAMA Intern Med. 2014 Apr;174(4):527-33. doi: 10.1001/jamainternmed.2013.14387. PMID 24515493
- [Background] West CP, Dyrbye LN, Erwin PJ, Shanafelt TD. Interventions to prevent and reduce physician burnout: a systematic review and meta-analysis. Lancet. 2016 Nov 5;388(10057):2272-2281. doi: 10.1016/S0140-6736(16)31279-X. Epub 2016 Sep 28. PMID 27692469
- [Background] Panagioti M, Panagopoulou E, Bower P, Lewith G, Kontopantelis E, Chew-Graham C, Dawson S, van Marwijk H, Geraghty K, Esmail A. Controlled Interventions to Reduce Burnout in Physicians: A Systematic Review and Meta-analysis. JAMA Intern Med. 2017 Feb 1;177(2):195-205. doi: 10.1001/jamainternmed.2016.7674. PMID 27918798